CLINICAL TRIAL: NCT03431571
Title: Use of the VisuMax Femtosecond Laser Lenticule Removal Procedure for the Correction of Hyperopia With or Without Astigmatism
Brief Title: Use of the VisuMax Femtosecond Laser Lenticule Removal Procedure for the Correction of Hyperopia
Acronym: V1601CI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Carl Zeiss Meditec AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V1601CI
Record Dates: First submitted 2018-01-26; First posted 2018-02-13 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Hypermetropia
Keywords: ReLEx; SMILE; Hyperopia; VisuMax; Small Incision Lenticule Extraction; Lenticule; Farsightedness
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): ReLEx SMILE treatment can be done binocular or monocular, no masking and randomization used, no control group
  Interventions: Procedure: ReLEx SMILE

INTERVENTIONS:
Procedure: ReLEx SMILE — the VisuMax femtosecond laser is used to cut a thin layer of corneal tissue that is removed through a small cut in the cornea

SUMMARY:
The correction of farsightedness using ReLEx SMILE for hyperopia is focus of this investigation. The objective is to evaluate the safety and effectiveness.

DETAILED DESCRIPTION:
The VisuMax laser keratome is an ophthalmic surgical femtosecond laser intended for use in patients requiring corneal incisions. The cutting action of the VisuMax laser keratome is achieved through precise individual micro-photodisruptions of tissue, created by tightly focused, ultra-short pulses, delivered through a disposable applanation lens while fixating the eye under a low vacuum. ReLEx SMILE combines state-of-the-art femtosecond laser technology of the VisuMax with high-precision lenticule extraction to provide minimally invasive refractive correction. It is distinguished by its flapless, minimally invasive laser correction. A refractive lenticule is created in the intact cornea, but removed via a small incision. The changed form of the cornea corrects the refraction error. ReLEx SMILE for myopia is a well-established treatment with extensive supporting published evidence for efficacy and safety. It is CE marked and available since 2011; more than 1 Million procedures have been performed worldwide. The correction of farsightedness using ReLEx SMILE for hyperopia is focus of this investigation and is therefore not yet CE marked.

ELIGIBILITY:
Inclusion Criteria:

* Normal corneal topography;
* Predicted post-operative keratometry ≤51 D;
* Contact lens wearers must stop wearing their contact lenses before baseline measurements according to local requirements of the clinic;
* Patients should be able to understand the patient information and willing to sign an informed consent;
* Patients should be willing to comply with all follow-up visits and the respective examinations;
* Patients with hyperopia or hyperopia with astigmatism (attempted correction: sphere up to +6.00D, cylinder up to 5.00D and maximum hyperopic meridian up to +7.00D);
* The corrected distance visual acuity should be 20/25 or better in each eye pre-operatively;
* A difference between cycloplegic and manifest refractions of ≤1.00 D spherical equivalent in the eye to be treated;

Exclusion Criteria:

* The patients presenting at least one of the characteristics as described for exclusion criteria in the documentation set of the VisuMax laser keratome ReLEx SMILE option.
* Mixed astigmatism
* Any impaired person (minors, pregnant or breast feeding women or persons incapable of giving consent) are definitely excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Corrected Distance Visual Acuity (CDVA) | 12 months
  CDVA in logMar

SECONDARY OUTCOMES:
side effects | 12 months
  distribution in percent
contrast sensitivity | 12 months
  contrast sensitivities for all spatial frequencies (3, 6, 12 and 18 cpd) in logMar
patient satisfaction (Quality of Vision Questionnaire) | 12 months
  Mean +/- standard deviation
manifest refractive astigmatism | 12 months
  Astigmatism in diopters [D]
spherical equivalent (SE) | 12 months
  SE in diopters [D]

CONTACTS AND LOCATIONS:
Overall Officials: Walter Sekundo, Principal Investigator — Uniklinikum Gießen Marburg
Locations (8):
- China (2):
  - University Medical Center Shanghai, Shanghai
  - Tianjin Eye Hospital, Heping District, Tianjin
- Gemini Eye Clinic, Zlín, Czechia
- University Medical Center CHRU Brest, Brest, France
- Germany (2):
  - Medical Center Heliosklinikum, Erfurt
  - University Medical Center Universitätsklinikum Gießen Marburg, Marburg
- Medical Center Nethradhama Superspeciality Eye Hospital, Bangalore, India
- London Vision Clinic, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No